CLINICAL TRIAL: NCT06931028
Title: A Randomized, Double-Blind, Placebo-Controlled Phase III Clinical Study to Assess the Efficacy and Safety of IBI362 in Chinese Subjects With Moderate-to-Severe Obstructive Sleep Apnea and BMI≥28 kg/m2 (GLORY-OSA)
Brief Title: A Study of IBI362 in Chinese Subjects With Obstructive Sleep Apnea and BMI≥28 kg/m2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIBI362E301
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Sleep Apnea; Obstructive; Obesity
MeSH Terms: conditions — Sleep Apnea Syndromes; Obesity | interventions — mazdutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Placebo Comparator): Participants receive placebo by subcutaneous (SC) injection once a week.
  Interventions: Other: placebo
- IBI362 (Experimental): ①2mg, SC, once a week* 4weeks; ②4mg, SC, once a week* 4weeks；③6mg, SC, once a week* 4weeks，9mg,SC,once a week* 36weeks
  Interventions: Drug: IBI362

INTERVENTIONS:
Other: placebo — placebo administered subcutaneously (SC) once a week.
  Arms: placebo
Drug: IBI362 — Once-weekly injections of gradually increased doses of IBI362
  Arms: IBI362

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase III clinical study to evaluate the efficacy and safety of IBI362 in subjects with moderate-to-severe obstructive sleep apnea (OSA) and a body mass index (BMI) ≥28 kg/m2. Subjects will be randomly assigned to IBI362 9 mg and placebo groups. All study treatment will be administered once-weekly and subcutaneously. The entire trial cycle includes a 4-week screening period, a 48-week double-blind treatment period, and a 12-week drug withdrawal follow-up period after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* For PAP s: Subjects who have received positive airway pressure (PAP) therapy for at least 3 consecutive months prior to screening and plan to continue PAP therapy during the study.
* For non-PAP s:Subjects who are unable or unwilling to undergo PAP therapy. PAP must not have been used for at least 4 weeks prior to screening.
* For all subjects:

  1. Age ≥18 years at the time of signing informed consent.
  2. Polysomnography (PSG) during screening shows an apnea-hypopnea index (AHI) ≥15 events/hour.
  3. Body mass index (BMI) ≥28.0 kg/m² at screening.

Exclusion Criteria:

For PAPs：

* Have personal or job-related responsibilities, or in the opinion of the investigator have any situation, that would make it unsafe to stop PAP therapy for 7 days prior to PSG testing during the course of the study
* Are unwilling to stop PAP therapy for 7 days prior to polysomnography (PSG) testing during the course of the study For all subjects：
* Have type 1 diabetes mellitus (T1DM) or type 2 diabetes mellitus (T2DM).
* Any previous or planned surgery for sleep apnea or major ear, nose or throat surgery, including tonsillectomy and adenoidectomy that still may affect breathing at time of baseline
* Have significant craniofacial abnormalities that may affect breathing at baseline
* Diagnosis of Obesity Hypoventilation Syndrome or daytime hypercapnia.
* Active device treatment of OSA other than PAP therapy (for example, dental appliance), or other treatment, that in the opinion of the investigator, may interfere with study outcomes, unless willing to stop treatment at baseline and throughout the study.
* Respiratory and neuromuscular diseases that could interfere with the results of the trial in the opinion of the investigator.
* Have achieved a >5% change in body weight through diet and exercise alone for at least 12 weeks prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2027-05-07 (Estimated); Study Completion 2027-06-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Apnea-Hypopnea Index (AHI) | Week 48
  AHI is defined as the average number of apnea and hypopnea events per hour of sleep, which is determined by polysomnography. The lower the value, the better, and the normal range is <5 events/hour.

SECONDARY OUTCOMES:
Percent Change from Baseline in Body Weight | Week 48
Change from Baseline in Systolic Blood Pressure (SBP) | Week 48
Percent Change from Baseline in Apnea-Hypopnea Index (AHI) | Week 48
  AHI is defined as the average number of apnea and hypopnea events per hour of sleep, which is determined by polysomnography. The lower the value, the better, and the normal range is <5 events/hour.
Percentage of Participants with ≥50% AHI Reduction from Baseline | Week 48
Percentage of Participants with AHI <5 or with AHI 5-14 with Epworth Sleepiness Scale (ESS) ≤10 | Week 48
Change from Baseline in Sleep Apnea-Specific Hypoxic Burden (SASHB) | Week 48
  SASHB is an indicator that quantifies the cumulative effect of hypoxia caused by apnea or hypopnea events during sleep. It is also calculated based on the results of polysomnography. It combines the severity, duration and frequency of hypoxia, and can more comprehensively reflect the systemic damage of hypoxia to the body. It is an important predictive factor for increased CVD risk. The lower the value, the better.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No